CLINICAL TRIAL: NCT00328146
Title: Re-operative Surgery in Children: A Technique for Sternal Re-Entry
Brief Title: Re-operative Surgery in Children:A Technique for Sternal Re-Entry
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-105
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; re-operative surgery
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation of Sternal Re-entry: All subjects.
  Interventions: Other: Observation of sternal reentry

INTERVENTIONS:
Other: Observation of sternal reentry — Observation of sternal reentry

SUMMARY:
Re-operative surgery in children is extremely challenging and injury to the underlying cardiac structures can occur during sternal re-entry. When institution of cardiopulmonary bypass is required in an emergency, there are often limited sites for peripheral cannulation. Injury to the heart can easily result in catastrophic complications and death.

DETAILED DESCRIPTION:
Background Re-operative surgery in children is extremely challenging and injury to the underlying cardiac structures can occur during sternal re-entry. When institution of cardiopulmonary bypass is required in an emergency, there are often limited sites for peripheral cannulation. Injury to the heart can easily result in catastrophic complications and death.

Methods This will be primarily a technique paper. The only clinical data points I am interested in are how many re-operative sternotomies we performed and on how many patients. I will also need to confirm that we did not have any complications due to cardiac injury while opening the sternum. I estimate about 450 patients.

Primary Aim: Present an effective technique for sternal re-entry in children

Secondary Aim: Present a zero incidence of complicated sternal re-entry over the past 5 years (February 1, 2001 through February 28, 2006) at Children's Healthcare of Atlanta, Egleston Hospital.

Inclusion / Exclusion Criteria Any child undergoing re-operative cardiac surgery through a midline sternotomy incision

ELIGIBILITY:
Inclusion Criteria:

* Any child undergoing re-operative cardiac surgery through a midline sternotomy incision

Exclusion Criteria:

* Those who do not fall under the above inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any child undergoing re-operative cardiac surgery through a midline sternotomy incision. This is a chart review.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2001-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Present an effective techniqe for sternal re-entry in children.

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States